CLINICAL TRIAL: NCT06262464
Title: The Efficacy of an OCD Prevention Programme for at Risk Adults: a Randomized Clinical Trial
Brief Title: An OCD Prevention Programme for at Risk Adults
Acronym: ØCD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Collaborators: Romanian National Authority for Scientific Research (Unknown)
Responsible Party: Principal Investigator, Roxana Cardos, Principal Investigator, Babes-Bolyai University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 17.361/ 07.12.2023
Record Dates: First submitted 2024-02-08; First posted 2024-02-16 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-03

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Risk; Prevention
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prevention (Experimental): 6 group, online sessions over two weeks. A prevention program using cognitive and behavioral strategies to reduce OCD risk factors and related symptoms.
  Interventions: Behavioral: Prevention
- Control (No Intervention): Treatment as Usual

INTERVENTIONS:
Behavioral: Prevention — A cognitive-behavioural prevention programme.
  Arms: Prevention

SUMMARY:
The main purpose of this randomised clinical trial is to test the efficacy of a prevention program for adult who are at risk of developing OCD, thus constituting a form of tertiary prevention.

DETAILED DESCRIPTION:
After being informed about the study and giving written informed consent, all eligible participants will be randomised into the experimental group or the control group (TAU). Participants will be blind to the group allocation.

The experimental group will undergo a two weeks OCD prevention program, consisting of three group sessions per week.

The control group will not receive any intervention.

Researchers will compare the experimental group to the control group to test wether the prevention programme is efficient in reducing OCD symptomatology.

ELIGIBILITY:
Inclusion Criteria:

- age over 18

Exclusion Criteria:

* clinically diagnosed OCD
* current psychiatric/psychotherapeutic treatment
* personality disorder diagnosis
* suicidal ideation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-02-09 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in OCD symptoms on the OCI-R after the intervention | Baseline and Week 2
  The OCI-R is a validated self-report instrument assessing OCD symptoms. Possible scores range from 0 to 72. Change = end of intervention score - baseline score
Change from baseline in depressive symptoms on the PHQ-9 after the intervention | Baseline and Week 2
  The PHQ-9 is a validated self-report instrument assessing depressive symptoms. Possible scores range from 0 to 27.
  Change = end of intervention score - baseline score
Change from baseline in anxiety symptoms on the GAD-7 after the intervention | Baseline and Week 2
  The GAD-7 is a validated self-report instrument assessing anxiety symptoms. Possible scores range from 0 to 21.
  Change = end of intervention score - baseline score

SECONDARY OUTCOMES:
Change from baseline in experiential avoidance on the EAQ after the intervention | Baseline and Week 2
  The EAQ is a validated self-report instrument assessing experiential avoidance. Possible scores range from 15 to 90.
  Change = end of intervention score - baseline score
Change from baseline in cognitive distortions on the OBQ-44 after the intervention | Baseline and Week 2
  The OBQ-44 is a validated self-report instrument assessing cognitive distortions in OCD. Possible scores range from 7 to 308.
  Change = end of intervention score - baseline score
Change from baseline in uncertainty intolerance on the IUS after the intervention | Baseline and Week 2
  The IUS is a validated self-report instrument assessing intolerance of uncertainty. Possible scores range from 27 to 135.
  Change = end of intervention score - baseline score
Change from baseline in resilience on the RSA after the intervention | Baseline and Week 2
  The RSA is a validated self-report instrument assessing resilience in adults. Possible scores range from 43 to 215.
  Change = end of intervention score - baseline score

OTHER OUTCOMES:
Change from baseline in life quality on the WHOQOL-BREF after the intervention | Baseline and Week 2
  The WHOQOL-BREF is a validated self-report instrument assessing life quality in adults.
  Change = end of intervention score - baseline score
Change from baseline in irrationality on the ATQ after the intervention | Baseline and Week 2
  The ABS-AV is a validated self-report instrument assessing irrationality in adults. Possible scores range from 24 to 120 Change = end of intervention score - baseline score
Change from baseline in global health on the GHQ-12 after the intervention | Baseline and Week 2
  The GHQ-12 is a validated self-report instrument assessing global health in adults.
  Possible scores range from 0 to 36. Change = end of intervention score - baseline score

CONTACTS AND LOCATIONS:
Overall Officials: Roxana Cardoș, PhD, Principal Investigator — Babeș-Bolyai University
Locations (1):
- Babes-Bolyai University, Faculty of Psychology and Educational Sciences, Department of Clinical Psychology and Psychotherapy, Cluj-Napoca, Romania, Romania

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The documents will be shared in March 2024

REFERENCES:
- [Derived] Cardos RAI, Dumitru EP, David OA. OCD: protocol for the development and evaluation of a cognitive-behavioral prevention program for obsessive-compulsive disorder. BMC Psychiatry. 2024 May 9;24(1):348. doi: 10.1186/s12888-024-05791-3. PMID 38724961